CLINICAL TRIAL: NCT02580188
Title: The Effect of Deep Neuromuscular Block on Surgical Condition During Laparoscopic Colorectal Surgery
Acronym: DEEPCOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, assistant proffesor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DNMBC-SNUBH
Record Dates: First submitted 2015-09-30; First posted 2015-10-20 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular blockade; Sugammadex; Laparoscopic surgery; Intra abdominal pressure alarm
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate block (No Intervention): Maintenance dose of 0.15-0.3 mg/kg/hr rocuronium as continuous infusion during surgery for the maintenance of train of four count 1-2 (moderate block). At the end of surgery neostigmine 50 ㎍/kg with glycopyrrolate 10 ㎍/kg are administered IV for reversal of neuromuscular block.
- Deep block (Experimental): Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium as continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium as continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block).
  Other Names: deep block
  Arms: Deep block

SUMMARY:
This study is a randomized, controlled, double-blinded, and parallel design study. A total 96 patients were randomized to receive a deep block or a moderate block scheduled for elective laparoscopic colorectal surgery. Investigators estimated the proportion of intra-abdominal pressure(IAP) alarm and surgical rating score.

DETAILED DESCRIPTION:
Patients >18 years of age with an america society of anesthesiologist classification of I or II who were scheduled to undergo elective laparoscopic colorectal surgery were included. The exclusion criteria were a history of neuromuscular, renal, or hepatic disease, a history of low abdominal surgery; treatment with drugs known to interfere with neuromuscular function. Patients were randomised to either the moderate or deep neuromuscular blockade group using Random Allocation Software (version 1.0). Premedication with intravenous midazolam at 0.03 mg/kg was performed in the reception area. In the operating room, routine monitoring was performed, including electrocardiography, non-invasive arterial pressure measurements, and pulse oximetry. Additionally, acceleromyography was applied to monitor the response of the corrugator supercilii muscle. Neuromuscular management and monitoring were performed according to the Good Clinical Research Practice guidelines. After the induction of anaesthesia with propofol and remifentanil using target-controlled infusers and before rocuronium administration, the TOF-Watch-SX was calibrated and stabilised; a 50-Hz tetanic stimulation was applied for 5 s, the TOF-Watch-SX was calibrated, and a series of train-of-four (TOF) measurements were documented for >2 min until a stable baseline was obtained (<5% variation in the TOF ratios). Next, intravenous rocuronium at 0.6 mg/kg was administered, and tracheal intubation was performed after confirmation of relaxation. Anesthesia was maintained with desflurane and target-controlled infusion of remifentanil while monitoring the bispectral index. A continuous dose of intravenous rocuronium (10-60 mg/hr) was used to maintain moderate (TOF count of 1 or 2) or deep (post-tetanic count [PTC] of 1 or 2) neuromuscular blockade. The IAP alarm(IAP>15mmHg) rate were checked. Any movement during the operation as reported by the surgeon or anaesthesiologist was recorded. At the end of the operation, the surgeon rated the surgical condition on a 5-point scale. Patients in the moderate group were reversed with neostigmine at 50 µg/kg and glycopyrrolate at 10 µg/kg at a TOF count of 1 or 2, and patients in the deep group were reversed with intravenous sugammadex at 4 mg/kg at PTC of 1 or 2. The time from administration of the reversal agents to a TOF ratio of 0.9 was recorded. Postoperative pain and opioid consumption were evaluated at 24, 48h postoperatively. Postoperative nausea and/or vomiting, dry mouth, were also evaluated at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade 1 or 2
* Scheduled for elective laparoscopic Colorectal surgery

Exclusion Criteria:

* Severe respiratory or cardiac disease
* Severe hepatic or renal function impairment
* On medications affecting neuromuscular function
* Known allergy to the drugs to be used
* Pregnant
* Malignant hyperthernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ah-Young Oh, MD.,Ph.D., Study Chair — Seoul national univ. BUNDANG hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group M: Maintenance dose of 0.15-0.3 mg/kg/hr rocuronium is continuous infusion during surgery for the maintenance of train of four count 1-2 (moderate block). At the end of surgery neostigmine 50 ㎍/kg with glycopyrrolate 10 ㎍/kg are administered IV for reversal of neuromuscular block.
- Group D: Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium is continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block
  sugammadex: Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium is continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block).
Period: Overall Study
Arm/Group | Group M | Group D
Started | 35 | 35
Completed | 32 | 32
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group M | Group D | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 14 | 11 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increased Intra-abdominal Pressure (IAP) Alarm as > 15 mmHg
Description: Intra-abdominal pressure was maintained at 12 mmHg during pneumoperitoneum(using the carbon dioxide gas insufflation) and the pressure alarm for IAP was set at < 15 mmHg.
  Intra-abdominal pressure is measured in a separate machine connected to a carbon dioxide gas injection line.
Time Frame: intraoperative, an averrage of 3 hour
Measure: Count of Participants; unit: Participants
Groups:
- Deep Block: Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium as continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block). At the end of surgery, sugammadex 4 mg/kg are administered IV for reversal of neuromuscular block
  sugammadex: Maintenance dose of 0.4-0.9 mg/kg/hr rocuronium is continuous infusion during surgery for the maintenance of post tetanic count 1-2 (deep block).
Arm/Group | Moderate Block | Deep Block
Number analyzed (Participants) | 32 | 32
Participants | 14 | 6

2. Other Pre Specified Outcome: Postoperative Pain is Evaluated by Verbal Numerical Rating Scale (VNRS, 0 = no Pain, 10 = the Severest Pain Imaginable)
Description: Postoperative pain is controlled by IV patient controlled analgesia using fentanyl. If patient complain of severe pain (VNRS score of 7 or more), additional analgesics can be used according to the attending physician.
Time Frame: 24hr after end of operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Moderate Block | Deep Block
Number analyzed (Participants) | 32 | 32
score on a scale | 4.5 [1 to 7] | 4 [0 to 8]

3. Other Pre Specified Outcome: Postoperative Pain is Evaluated by Verbal Numerical Rating Scale (VNRS, 0 = no Pain, 10 = the Severest Pain Imaginable)
Description: as for outcome 2
Time Frame: 48hr after end of operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Moderate Block | Deep Block
Number analyzed (Participants) | 32 | 32
score on a scale | 3 [0 to 8] | 2 [0 to 7]

ADVERSE EVENTS:
Arm/Group | Group M | Group D
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No